CLINICAL TRIAL: NCT00389649
Title: Effect of Chronic Changes in Heart Rate on Congestive Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Stephen Gottlieb, Professor o Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H-20887
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Results first posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-11

CONDITIONS: Heart Failure, Congestive
Keywords: congestive heart failure; pacemaker; heart rate
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- HR=60 (Active Comparator): Pacemaker set at 60
  Interventions: Device: heart rate setting
- HR=75 (Active Comparator): Pacemaker set at 75
  Interventions: Device: heart rate setting
- HR=90 (Active Comparator): Pacemaker set at 90
  Interventions: Device: heart rate setting

INTERVENTIONS:
Device: heart rate setting

SUMMARY:
This will be a double blind randomized crossover study of patients with congestive heart failure and a heart rate dependent upon a permanent pacemaker. Thus, at all times the heart rate can be maintained at a set rate by adjusting the settings of the pacemaker. Acute and chronic effects of heart rates of 60, 75, and 90 beats per minute will be evaluated. The effect of heart rate will be determined by measuring ejection fraction by nuclear ventriculography, six minute walk distance, and peak oxygen consumption on a maximal exercise test.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, cross-over study of patients with congestive heart failure and a heart rate dependent on a permanent pacemaker. Thus, at all times the heart rate can be maintained at a set rate by adjusting the settings of the pacemaker. Acute and chronic effects of heart rates of 60, 75, and 90 beats per minute will be evaluated by primarily comparing cardiopulmonary exercise tests and radionuclide ventriculography scans.

Inclusion Criteria:

Patients must have symptomatic congestive heart failure, NYHA Class II to IV symptoms and an ejection fraction < 40% by nuclear ventriculography within the previous 6 months. Patients must be stable with no change in dosage on conventional therapy (including digoxin, diuretics, ACE inhibitors, hydralazine, nitrates, angiotensin II receptor blockers and/or beta blocker) for at least 4 weeks. Because only heart rate is being evaluated, stable treatment with beta blockade should not prevent evaluation of the effects of changing heart rate.

Patients must have an intrinsic cardiac rate < 60 beats per minute and a functioning permanent pacemaker.

Exclusion Criteria:

1. active alcohol or illicit drug use
2. myocardial infarction or unstable angina within the previous 3 months
3. obstructive valvular disease
4. exercise induced sustained arrhythmias or symptomatic myocardial ischemia
5. pregnancy
6. psychiatric disorder
7. non-compliance with medical regimen

Assessment for eligibility:

Patients who appear eligible based upon the prior inclusion and exclusion criteria will be further evaluated for eligibility as follows:

After signing a consent form but prior to randomization and enrollment, the pacemaker rate will be set at 60 and then a 24 hour assessment by Holter monitor will be obtained. Patients will be eligible for the study if they are paced at least 75% of the time. For rate responsive pacemakers, the pacemaker will be set at a lower rate of 60 and an upper rate of 80. Patients will need to be paced at a rate of 60 beats per minute at least 75% of the time for these patients as well.

A symptom limited maximal exercise tolerance with measurement of peak oxygen consumption (VO2) will be performed to assess patient's maximal aerobic capacity. The Naughton protocol will be used. Exercise will continue until limiting symptoms are present, but will be stopped if patient develops sustained arrhythmia, cyanosis, dizziness, decrease in blood pressure or an ataxic gait. Patients who develop angina or claudication limiting exercise capacity will be excluded from further evaluation or participation. Peak oxygen consumption on this test must be < 20 ml/kg/min for a patient to be eligible for this study.

Chronic Study

Randomization:

This study will be a three period crossover study. Patients initially will be randomly assigned to be paced at a rate of 60, 75, or 90 BPM for 2 consecutive months. Patients with rate responsive pacemakers will be set at an upper limit of 20 beats above their assigned rate. At the end of this period, patients will have end point measurements obtained and then will be randomized to one of the other heart rates for another 2 consecutive months. Following repeat end point measurements at the end of this period, patients will then be randomized to the final heart rate for 2 consecutive months with repeat measurements at the end.

End Point Measurements:

The following tests will be done at the end of each of the three two month periods to assess the effect of heart rate on ventricular function, functional status and exercise capacity.

1. Nuclear ventriculography (MUGA): Equilibrium gated blood pool will be completed according to standard protocol, under the supervision of Dr. Eliot Siegel. Ejection fraction will be calculated.
2. Six minute walk: All patients will have their submaximal exercise capacity evaluated by a 6 minute walk. This test is performed on a 100 foot hallway. Patients are instructed to walk from end to end repeatedly at a comfortable pace while attempting to cover as much ground as possible. After 6 minutes the distance covered is measured to the nearest foot.
3. Maximal exercise tolerance and peak oxygen consumption: This will be assessed in all patients at baseline and at the end of each 2 month period. Patients will be exercised to exhaustion on a motorized treadmill using a Naughton Protocol. Heart rate and rhythm will be monitored continuously while blood pressure will be measured every 2 minutes. Oxygen consumption, C02 production and respiratory quotient will be calculated every 20 seconds using breath by breath analysis.

Acute Studies Effect of Heart Rate on Ejection Fraction Acute studies will be performed to help differentiate the effect of changes in heart rate on left ventricular ejection fraction from changes in cardiac performance and contractility. Acutely, ejection fraction might change because of alterations in preload and afterload, which might not reflect the long term effects on contractility.

At the end of the first 2 month period, the patient will have nuclear ventriculography (as detailed above) to evaluate ejection fraction. At that time the pacemaker rate will be changed in a random manner to the two other heart rates. Ten minutes after each adjustment, an ejection fraction will be calculated.

Effect of Heart Rate on Exercise Performance:

The purpose of this study is to look at the acute effect of changes in heart rate on exercise performance. This will differentiate exercise effects induced by the change in heart rate on contractility from the acute effects of changing heart rate. Twenty four hours following randomization of patients to the first heart rate, they will have an exercise tolerance test. As previously indicated, the effect of a chronic change in heart rate ill be evaluated following each 2 month period. Subsequently, when patients are crossed over to another heart rate, they will have an exercise tolerance test 24 hours later. This will follow the chronic exercise test of the previous period by at least 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have symptomatic congestive heart failure, NYHA Class II to IV symptoms and an ejection fraction < 40% by nuclear ventriculography within the previous 6 months. Patients must be stable with no change in dosage on conventional therapy (including digoxin, diuretics, ACE inhibitors, hydralazine, nitrates, angiotensin II receptor blockers and/or beta blocker) for at least 4 weeks

Exclusion Criteria:

* active alcohol or illicit drug use
* myocardial infarction or unstable angina within the previous 3 months
* obstructive valvular disease
* exercise induced sustained arrhythmias or symptomatic myocardial ischemia
* pregnancy
* psychiatric disorder
* non-compliance with medical regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2001-11; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gottlieb, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 60, 75, 90: Pacemaker set at HR=60 for 1 month, 75 for 1 month and 90 for 1 month
- 60, 90, 75: HR=60 for 1 month, 90 for 1 month and 75 for 1 month
- 75, 60, 90: HR=75 for 1 month, 60 for 1 month and 90 for 1 month
- 75, 90, 60: HR=75 for 1 month, 90 for 1 month and 60 for 1 month
- 90, 60, 75: HR=90 for 1 month, 60 for 1 month and 75 for 1 month
- 90, 75, 60: HR=90 for 1 month, 75 for 1 month and 60 for 1 month
Period: Overall Study
Arm/Group | 60, 75, 90 | 60, 90, 75 | 75, 60, 90 | 75, 90, 60 | 90, 60, 75 | 90, 75, 60
Started | 2 | 2 | 3 | 2 | 2 | 2
Completed | 2 | 2 | 3 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 60,75,90: HR set at 60 for 1 month, then 75, then 90
- 60,90,75: HR set at 60 for 1 month, then 90, then 60
- 75, 60, 90: HR set at 75 for 1 month, then 60, then 90
- 75, 90, 60: HR set at 75 for 1 month, then 90, then 60
- 90, 60, 75: HR set at 90 for 1 month, then 60, then 75
- 90, 75,60: HR set at 90 for 1 month, then 75, then 60
- Total: Total of all reporting groups
Arm/Group | 60,75,90 | 60,90,75 | 75, 60, 90 | 75, 90, 60 | 90, 60, 75 | 90, 75,60 | Total
Number analyzed (Participants) | 2 | 2 | 3 | 2 | 2 | 2 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 1 | 0 | 0 | 5
  >=65 years | 1 | 0 | 2 | 1 | 2 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 1 | 0 | 0 | 3
  Male | 2 | 1 | 2 | 1 | 2 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Ejection Fraction
Description: Ejection fraction as measured by nuclear ventriculography
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: % of blood ejected with each beat
Groups:
- HR=60: Pacemaker set at 60
  heart rate setting
- HR=75: Pacemaker set at 75
  heart rate setting
- HR=90: Pacemaker set at 90
  heart rate setting
Arm/Group | HR=60 | HR=75 | HR=90
Number analyzed (Participants) | 13 | 13 | 13
% of blood ejected with each beat | 33 (6) | 30 (6) | 25 (6)

2. Secondary Outcome: Peak Oxygen Consumption
Description: Patients were exercised to exhaustion on a motorized treadmill using a modified Naughton protocol. Oxygen consumption, was calculated
Time Frame: 2 months
Population: 3 patients were unable to have peak oxygen consumption assessed at all 3 time points
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | HR=60 | HR=75 | HR=90
Number analyzed (Participants) | 10 | 10 | 10
ml/kg/min | 11.0 (2.4) | 11.3 (2.9) | 9.5 (2.9)

3. Secondary Outcome: Distance Traveled During a 6 Minute Walk
Description: Patients had submaximal exercise capacity evaluated by a 6-minute walk. This test was performed on a 100-foot hallway. Patients were instructed to walk from end to end repeatedly at a comfortable pace while attempting to cover as much ground as possible. After 6 minutes, the distance covered was measured to the nearest foot.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | HR=60 | HR=75 | HR=90
Number analyzed (Participants) | 12 | 12 | 12
feet | 938 (293) | 996 (260) | 888 (284)

ADVERSE EVENTS:
Arm/Group | HR=60 | HR=75 | HR=90
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No